CLINICAL TRIAL: NCT06058403
Title: The Impact of Canola Protein Processing on Postprandial Plasma Amino Acid Responses in Vivo in Young Females
Brief Title: Impact of Canola Protein Processing on Plasma Amino Acid Responses
Acronym: CANOLAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: DSM Food Specialties (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL83369.068.23 / METC 23-025
Record Dates: First submitted 2023-09-05; First posted 2023-09-28 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Protein Metabolism Disorder
Keywords: Dietary protein; Plant protein; Protein processing; Protein digestion
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-blind, cross-over intervention trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Native canola protein (Experimental): 20g of canola protein
  Interventions: Dietary Supplement: 20g native canola protein drink ingestion
- Processed canola protein #1 (Experimental): 20g of processed canola #1
  Interventions: Dietary Supplement: 20g processed canola protein #1 drink ingestion
- Processed canola protein #2 (Experimental): 20g of processed canola #2
  Interventions: Dietary Supplement: 20g processed canola protein #2 drink ingestion
- Whey protein (Active Comparator): 20g of whey protein
  Interventions: Dietary Supplement: 20g whey protein drink ingestion

INTERVENTIONS:
Dietary Supplement: 20g whey protein drink ingestion — Ingestion of a 300 mL drink containing 20g whey protein
  Other Names: Supplement
  Arms: Whey protein
Dietary Supplement: 20g native canola protein drink ingestion — Ingestion of a 300 mL drink containing 20g native canola protein
  Other Names: Supplement
  Arms: Native canola protein
Dietary Supplement: 20g processed canola protein #1 drink ingestion — Ingestion of a 300 mL drink containing 20g processed canola protein #1
  Other Names: Supplement
  Arms: Processed canola protein #1
Dietary Supplement: 20g processed canola protein #2 drink ingestion — Ingestion of a 300 mL drink containing 20g processed canola protein #2
  Other Names: Supplement
  Arms: Processed canola protein #2

SUMMARY:
Muscle tissue consists of proteins. These proteins are built up of small building blocks: amino acids. By consuming enough protein through the diet, the body is provided with enough amino acids to facilitate muscle protein building. Providing the growing world population with sufficient animal-derived protein is a challenge. Plant proteins can be produced on a more sustainable commercial scale than conventional animal-derived proteins and therefore can contribute to feeding our future population. Canola protein is a protein that is derived from rapeseed. The composition of canola seems to be comparable to that of other high-quality animal based protein sources. However, the collection of canola protein from rapeseed occurs in a special way. These treatment processes might affect canola protein digestion. The goal of this study is to investigate the most optimal way of canola protein processing on blood plasma amino acid responses.

Primary objective: To assess the impact of canola protein processing on 5h postprandial plasma total amino acid incremental area under the curve (iAUC) in vivo in healthy young females.

Hypothesis: it is hypothesized that the ingestion of 20g processed canola will result in greater 5h postprandial plasma total amino acid iAUC in vivo in healthy young females, when compared to the ingestion of 20g native canola protein isolate.

DETAILED DESCRIPTION:
To assess whether volunteers are eligible to participate in this study, the investigator will invite them to the University for a screening. At the start of the screening session, the entire experimental trial will be explained, and any potential questions will be answered. Thereafter, the volunteers are asked to read, fill out, and sign the informed consent form. After signing the informed consent form, the participant's eligibility will be assessed based on the in- and exclusion criteria. To further asses their eligibility, participants will be asked to fill out a medical questionnaire to assess their general health, use of medication, habitual food intake, and physical activity. Next, blood pressure will be assessed. Body mass (with accuracy of 0.1 kg) and height (with accuracy of 0.01 m) will be determined. The screening sessions will take place in the morning and participants are instructed to not have any breakfast in the morning in order to avoid perturbations in body weight and possibly in the DEXA scan. In the event of an unexpected medical finding during the screening, subjects will always be notified. If a subject does not want to receive this notification, she cannot participate in the study. When the screening is successfully performed, the test days will be scheduled. Protein and amino acid metabolism in women can be influenced by the menstrual cycle. Therefore, the experimental test days will be standardized in a specific period of the menstrual cycle. The test days will be planned in the first 10 days after the start of the menses (day 1 of the follicular phase), when hormones levels (i.e., estrogen) are low. In practice, this means that the test days will be planned based on the subjects' menstrual cycle. Therefore, 2 test days can be performed within 1 menstrual cycle (allowing 2 days between test days for standardization) and further test days will be planned approximately 28 days thereafter. This allows the investigators to finish testing for a single participant within a relatively short time frame while still taking the menstrual cycle and accompanying hormonal influences into consideration. A similar approach was used in our lab in previous studies that included young healthy women (METC17-3-047 & METC19-087). Throughout the study period, participants will also undergo a fasted Dual Energy X-ray Absorptiometry (DEXA) scan to assess body composition. A DEXA scan is a simple, non-invasive procedure. At the beginning of the procedure, subjects will be asked to lie down on a scanning table wearing underwear and they need to remain motionless during the measurements. As the scanner moves, a dual energy beam passes through the targeted skeletal muscle section and is measured by a detector. This procedure takes approximately 3 minutes. The DEXA-scan provides valuable insight in participants' body composition, with minimal radiation burden.

When the screening is successfully performed, the test day will be scheduled. In order to prevent major impact from the menstrual cycle on the measurements of protein metabolism, the test day will be scheduled to take place in the first 10 days of the follicular phase.

Each subject will participate in 4 experimental test days lasting ~5h. Subjects will be instructed to arrive at the university at 8:45 AM in an overnight fasted and rested state, meaning that participants are not allowed to eat and drink (except for water) from 22:00 the night prior to the experimental trial. They will be instructed to come to the university by car or public transportation. After the subjects arrive at the University, subjects will rest in a seated position and a Teflon catheter will be inserted in a heated dorsal hand vein and placed in a hot-box (60°C) for arterialized blood sampling. A baseline blood sample (Serum + plasma = 20 mL) will be collected at t=0 min to determine the amino acid concentrations prior to the intervention.

Then, subjects will ingest the assigned drink (20g native canola protein, 20g processed canola protein #1, 20g processed canola protein #2, or 20g whey protein). Subjects will be instructed to consume the drink within ~5 min. Upon drink ingestion, the stopwatch will be started (t= 0 min), and arterialized blood samples (10mL) will be collected at t = 15, 30, 45, 60, 90, 120, 180, 240, and 300 min. During the entire experimental test day, the hand with the dorsal hand catheter will be pre-heated for 10 minutes prior to every blood draw in a hot box at 60°C to increase blood flow. This makes it easier to collect blood and minimizes nutrient exchange from blood into other tissues. Therefore, it allows the investigators to collect nutrient-rich (arterialized) blood from a vein.

In total 10 times blood samples will be taken during the test day, the first sample that will be collected will be 20mL and subsequent samples will be 10mL, making a total of 110mL.

Additionally, gastro-intestinal (GI) symptoms will be assessed at t = 0, 30, and 180 minutes and palatability at t = 15 min by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Aged between 18 and 35 y inclusive
* BMI between 18.5 and 30 kg/m2

Exclusion Criteria:

* Intolerant to milk lactose
* Allergic to milk protein / products
* Mustard allergy
* Vegan lifestyle
* Participating in a structured (progressive) exercise program
* Smoking regularly
* Diagnosed GI tract disorders or diseases
* Diagnosed musculoskeletal disorders
* Diagnosed metabolic disorders (e.g., diabetes)
* Hypertension (blood pressure above 140/90 mmHg)
* Donated blood 2 months prior to test day
* Pregnant
* Using third generation oral contraceptives
* Use of any medications known to affect protein metabolism (i.e., corticosteroids, non-steroidal anti-inflammatories).
* Chronic use of gastric acid suppressing medication as this impairs protein digestion (i.e., proton pump inhibitors, H2-antagonists)
* People with Phenylketonuria

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Total amino acid availability | 0 - 5 hours after drink ingestion
  The total amino acid availability is expressed as the incremental area under the curve (iAUC)

SECONDARY OUTCOMES:
Postprandial plasma total amino acid concentrations | 0 - 5 hours after drink ingestion
  The total plasma amino acid concentrations from the sum of the individual amino acids
Postprandial plasma individual amino acid concentrations | 0 - 5 hours after drink ingestion
  The plasma amino acid concentrations of the individual amino acids
Peak plasma amino acid concentrations | 0 - 5 hours after drink ingestion
  The maximal plasma amino acid concentrations
Time to peak plasma amino acid concentrations | 0 - 5 hours after drink ingestion
  The time to reach maximal plasma amino acid concentrations
iAUC essential amino acids concentrations | 0 - 5 hours after drink ingestion
  Essential amino acid availability expressed as incremental area under the curve (iAUC)
iAUC non-essential amino acid concentrations | 0 - 5 hours after drink ingestion
  non-essential amino acid availability expressed as incremental area under the curve (iAUC)
Plasma insulin concentrations | 0 - 5 hours after drink ingestion
  Postprandial plasma insulin concentrations

OTHER OUTCOMES:
Age in years | Baseline at screening
  Age in years reported by participants
Bodymass in kg | Baseline at screening
  Scale
Height in m | Baseline at screening
  Statiometer
BMI in kg/m^2 | Baseline at screening
  calculated from height and body mass
Whole body lean mass in kilograms | Up to 3 months after inclusion
  DEXA
Appendicular lean mass | Up to 3 months after inclusion
  DEXA
Bodyfat% | Up to 3 months after inclusion
  DEXA
Dietary energy intake | Two days prior to first experimental trial day
  Assessed by written dietary intake records
Dietary protein intake | Two days prior to first experimental trial day
  Assessed by written dietary intake records
Dietary fat intake | Two days prior to first experimental trial day
  Assessed by written dietary intake records
Dietary carbohydrate intake | Two days prior to first experimental trial day
  Assessed by written dietary intake records
Drink palatability | On experimental trial day directly after drink ingestion
  Assessed by visual analogue scale after drink ingestion. Higher score means better taste (scoring 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boot N, Hermans WJH, Warnke I, Overman A, van Kranenburg JMX, Senden JM, Verdijk LB, van Loon LJC. Evaluation of processing of canola protein isolate on postprandial plasma amino acid profiles in healthy, young females. Amino Acids. 2025 Oct 17;57(1):50. doi: 10.1007/s00726-025-03482-1. PMID 41107640